CLINICAL TRIAL: NCT00268034
Title: Left Ventricular Aneurysms in Children
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 04-073
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Disorders
Keywords: pediatric; cardiac; aneurysms; left ventricular aneurysms; surgical repair for LV aneurysms
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Aneurysm

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
Collect data to support "standard of care possibility" of extracardiac repair with closure of intracavitary communication and plication of the aneurysm as probably safest surgical repair for left ventricular aneurysms.

DETAILED DESCRIPTION:
Ventricular aneurysms in the pediatric population are rare and no standardized method of treatment exists.

We plan on reviewing five patient charts between the dates of 6.30.02 and 6.30.04 as to causes of aneurysms. The patient charts selected will be in the following "aneurysm categories":

Mostly occur after:

Ross/Ross-Konno procedures modified Rastelli-type interventricular tunnels repeated resections of subaortic stenosis and possibly after: myocardial ischemia trauma drainage of abscess in infective endocarditis progressive herniation of endocardium mostly located: in LV outflow tract

We plan on collecting echocardiograms and / or cardiac catheterizations data in order to confirm the diagnosis of an aneurysm. We will also collect the following information:

* Procedures including the dates performed
* Medications
* Physical Exam Findings
* Weight
* Gestational Age
* Outcome

ELIGIBILITY:
Inclusion Criteria:

* aneurysms between 6.30.2002 and 6.30.2004

Exclusion Criteria:

* those children who do no meet inclusion criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5
Dates: Start 2002-06

CONTACTS AND LOCATIONS:
Overall Officials: Kirk R Kanter, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States